CLINICAL TRIAL: NCT05679206
Title: Association Between Preeclampsia, Antiphospholipid Syndrome and Postpartum Pulmonary Artery Pressure, Systemic Arterial Pressure and Cardiovascular Function.
Brief Title: Antiphospholipid Syndrome and Postpartum Pulmonary Artery Pressure
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Emrush Rexhaj, Head of Hypertension, Principal Investigator, Insel Gruppe AG, University Hospital Bern
Other Study IDs: 2022-01957
Record Dates: First submitted 2022-12-21; First posted 2023-01-10 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Pre-Eclampsia; Complicating Pregnancy; Antiphospholipid Syndrome in Pregnancy; Pulmonary Hypertension
Keywords: Pre-Eclampsia; Antiphospholipid Syndrome in Pregnancy; Pulmonary Hypertension
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications; Hypertension, Pulmonary | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preeclampsia and obstetric Antiphospholipid Syndrome: Women in this group wil be followed during 3 years. Echocardiography images, 24-hour ambulatory blood pressure monitoring will be collected.
  Interventions: Diagnostic Test: Echocardiography images; Diagnostic Test: 24-hour ambulatory blood pressure monitoring
- Preeclampsia without obstetric Antiphospholipid Syndrome: Women in this group wil be followed during 3 years. Echocardiography images, 24-hour ambulatory blood pressure monitoring will be collected.
  Interventions: Diagnostic Test: Echocardiography images; Diagnostic Test: 24-hour ambulatory blood pressure monitoring

INTERVENTIONS:
Diagnostic Test: Echocardiography images — Transthoracic echocardiographic (Vivid E95) performed in all included patients between three months and three years after delivery.
  * Left ventricular ejection fraction,
  * Left ventricular mass index,
  * Septal and lateral mitral annular E-wave velocity assessed by tissue Doppler,
  * Tricuspid annular plane systolic excursion,
  * Left atrial volume index,
  * Right ventricle to right atrium (RV/RA) gradient
Diagnostic Test: 24-hour ambulatory blood pressure monitoring — Twenty-four-hour ABPM performed between three months and three years after delivery using validated recorders (Spacelabs model 90217, USA)

SUMMARY:
The primary goal of this observational study is to learn about postpartum pulmonary artery pressure in women who suffered from Preeclampsia and Antiphospholipid Syndrome.

The main question it aims to answer is whether the conjunction of preeclampsia with obstetric antiphospholipid syndrome significantly foster the development of long-lasting pulmonary hypertension.

Only participants who suffered from preeclampsia during pregnancy will be followed for a period up to 3 years postpartum. Researchers will compare women with or without obstetric antiphospholipid syndrome.

DETAILED DESCRIPTION:
Preeclampsia (PE), a multisystem disease affecting 2-8% of all pregnancies is a major cause of mother and child mortality and morbidity worldwide. On the long term, women who suffered from PE during pregnancy are prone to develop various cardiovascular diseases including arterial hypertension, heart failure, aortic stenosis, mitral regurgitation and atrial fibrillation.

In an effort to prevent or early detect any potential cardiovascular complications in this population, the investigators implemented in Inselspital, 6 years ago, a join consultation between cardiologist and obstetrician. Since 2016, a roughly 100 women/year have been followed at this consultation. As part of this follow-up, in addition to a clinical examination, echocardiography, blood sampling and 24h ambulatory blood pressure monitoring were performed. To the best of the investigators knowledge, this represent the first cohort of this kind in Switzerland. Therefore, it offers a unique opportunity to study the effect of PE on the long term cardiovascular phenotype.

Although the majority of PE are of unknown origin a fraction is due to an autoimmune disease, the Antiphospholipid Syndrome (APS). APS is known to triple the risk of developing PE and is found in up to 20% in women with the most severe forms of PE. There are two distinguished entities of APS, one associated with vascular complications (vascular APS) and one associated with adverse pregnancy outcomes (obstetric APS (oAPS)). In the former form, the prevalence of pulmonary hypertension has been reported to be between 2% and 17% (incidence in the general population ~ 1/100'000) but remain unknown in oAPS. This is of prime importance as pulmonary arterial hypertension is a rare disease with elevated mortality and limited treatment availability. Furthermore, for unknown raison, women have up to seven times the risk of men to develop PH. Here, the investigators hypothesize that oAPS could be an unrecognized risk factor for the development of PH in women.

In patients who suffered from PE, epidemiological studies shown that the risk for developing arterial hypertension, stroke or heart failure is 2-4 fold higher. But structured follow-up to better target this population is missing. Our established interdisciplinary consultation offer a unique possibility to better understand the link between PE and cardiovascular outcomes later in life. Therefore, the investigators further aimed in this study, first to assess the prevalence of the above mentioned cardiovascular outcomes, and second, to establish prediction models, for example for the development of arterial hypertension in patient that suffered from PE.

The primary objective of this study is to compare the postpartum pulmonary arterial pressure measured non-invasively by echocardiography in women after PE with or without oAPS by collecting routine data for the analysis.The secondary objective is to compare the right and left cardiac function using echocardiography images and the systemic blood pressure between both groups by collecting routine data for the analysis. Further, the investigators aimed to assess the prevalence of arterial hypertension in this population, 3 years postpartum and establish a prediction model of the development of arterial hypertension by collecting routine data for the analysis.

The investigators are planning a single center retrospective and prospective study where routine data is collected to evaluate the objectives described above. In particular, demographic, biophysical as well as echocardiographic parameters of all the patients whose pregnancies were complicated by preeclampsia, and were or will be referred after delivery to our outpatient clinic will be collected and analyzed. All consenting patients (see chapter 9) followed between 2016 and 2025 will be enrolled. All data will be collected during a period ranging from 2016 to 2028 encompassing the first patient enrolment in 2016 and the end of the 3 years routine follow-up of the last patient enrolled in 2025.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 16 years.
* Consent or waiver of consent according Chapter 9
* Preeclampsia

Defined as:

• New onset hypertension (blood pressure >140/90mmHg on multiple occasions after 20 weeks of gestation)

In combination with new onset of 1 or more of the following:

* Proteinuria (urine protein >300mg /24h or 2+ or higher in dipstick on multiple occasions)
* Platelet count <100,000/microL,
* Serum creatinine >97.2 micromol/L,
* Liver transaminases at least twice the upper limit of the normal concentrations,
* Pulmonary edema,
* New-onset and persistent headache,
* Visual symptoms. -Postnatal follow up at the obstetrical and cardiology clinic, Inselspital Bern, Switzerland.

Exclusion Criteria:

* Age: < 16 years
* Incomplete or ambiguous data: if data confirming the eligibility criteria or data to analyze the primary endpoint is not fully available or despite efforts assessed as significantly ambiguous, the data set will be excluded from analyses, since no analysis is possible

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will retrospectively and prospectively study a cohort of PE patient followed at our interdisciplinary postpartum consultation. Informed consent was/will be obtained by means of a general consent. Only for the analysis relevant clinical data (i.e. Echocardiography, ABPM and blood sampling results) will be extracted from the patient files and encoded (according Swissethics guideline) for further analysis.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in systolic pulmonary artery pressure | three months and three years after delivery
  Right ventricle to right atrium (RV/RA) gradient will be mesured using echocardiography

SECONDARY OUTCOMES:
Changes in systemic arterial blood pressure | three months and three years after delivery
  Twenty-four-hour ambulatory blood pressure monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Emrush Rexhaj, MD, Principal Investigator — Insel Gruppe AG, Inselspital, Bern
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benschop L, Duvekot JJ, Roeters van Lennep JE. Future risk of cardiovascular disease risk factors and events in women after a hypertensive disorder of pregnancy. Heart. 2019 Aug;105(16):1273-1278. doi: 10.1136/heartjnl-2018-313453. Epub 2019 Jun 7. PMID 31175138
- [Background] Brown MA, Magee LA, Kenny LC, Karumanchi SA, McCarthy FP, Saito S, Hall DR, Warren CE, Adoyi G, Ishaku S; International Society for the Study of Hypertension in Pregnancy (ISSHP). The hypertensive disorders of pregnancy: ISSHP classification, diagnosis & management recommendations for international practice. Pregnancy Hypertens. 2018 Jul;13:291-310. doi: 10.1016/j.preghy.2018.05.004. Epub 2018 May 24. No abstract available. PMID 29803330
- [Background] Heilmann L, Schorsch M, Hahn T, Fareed J. Antiphospholipid syndrome and pre-eclampsia. Semin Thromb Hemost. 2011 Mar;37(2):141-5. doi: 10.1055/s-0030-1270341. Epub 2011 Mar 2. PMID 21370215
- [Background] Honigberg MC, Zekavat SM, Aragam K, Klarin D, Bhatt DL, Scott NS, Peloso GM, Natarajan P. Long-Term Cardiovascular Risk in Women With Hypertension During Pregnancy. J Am Coll Cardiol. 2019 Dec 3;74(22):2743-2754. doi: 10.1016/j.jacc.2019.09.052. Epub 2019 Nov 11. PMID 31727424
- [Background] Leon LJ, McCarthy FP, Direk K, Gonzalez-Izquierdo A, Prieto-Merino D, Casas JP, Chappell L. Preeclampsia and Cardiovascular Disease in a Large UK Pregnancy Cohort of Linked Electronic Health Records: A CALIBER Study. Circulation. 2019 Sep 24;140(13):1050-1060. doi: 10.1161/CIRCULATIONAHA.118.038080. Epub 2019 Sep 23. PMID 31545680
- [Background] Olie V, Moutengou E, Grave C, Deneux-Tharaux C, Regnault N, Kretz S, Gabet A, Mounier-Vehier C, Tsatsaris V, Plu-Bureau G, Blacher J. Prevalence of hypertensive disorders during pregnancy in France (2010-2018): The Nationwide CONCEPTION Study. J Clin Hypertens (Greenwich). 2021 Jul;23(7):1344-1353. doi: 10.1111/jch.14254. Epub 2021 May 27. PMID 34042277
- [Background] Rana S, Lemoine E, Granger JP, Karumanchi SA. Preeclampsia: Pathophysiology, Challenges, and Perspectives. Circ Res. 2019 Mar 29;124(7):1094-1112. doi: 10.1161/CIRCRESAHA.118.313276. PMID 30920918